CLINICAL TRIAL: NCT05789238
Title: Development of Online Store for Testing Regulatory Food and Nutrition Policies in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-2129
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-04

CONDITIONS: Dietary Habits
Keywords: front-of-package labels; ANVISA; PAHO
MeSH Terms: conditions — Feeding Behavior | interventions — Pan American Health Organization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No labels for products high in added sugar, saturated fat, or sodium
- ANVISA (Experimental): Levels of added sugars, saturated fat, and sodium, if exceeded according to the Brazil Nutrient Profile Model, will require the magnifying glass FOPL below on the front of the package for either solid food or liquid food.
  Interventions: Behavioral: ANVISA
- PAHO (Experimental): PAHO Model is not based on thresholds (cut-off limits), but by percentage of regulated nutrient values in total calories amount and by NOVA categories. Therefore, the Brazil team has classified products from the dataset into NOVA categories and created calculations to apply the PAHO model to PdeA products.
  Interventions: Behavioral: PAHO

INTERVENTIONS:
Behavioral: ANVISA — Products carrying front-of-package labels based on Brazil's Health Regulatory Agency (ANVISA's) nutrient profile model
  Arms: ANVISA
Behavioral: PAHO — Products carrying front-of-package labels based on the Pan-American Health Organization (PAHO's) nutrient profile model
  Arms: PAHO

SUMMARY:
The purpose of this randomized controlled trial is to assess the impact of different nutrient profiles for magnifying glass front-of-package labels (FOPLs) on consumer choices in an online grocery store. Participants will be adults residing in Brazil recruited through a survey research firm. Participants will be randomly assigned to one of three shopping environments in an online grocery store. Participants will complete a shopping task (selecting items from a pre-specified shopping list) in the online grocery store. After completing the shopping task, participants will be rerouted to a computer survey. The survey will include standard behavior and label perception questions, as well as demographic items.

DETAILED DESCRIPTION:
Among noncommunicable disease, cardiovascular-related diseases are the leading cause of death worldwide and contribute to almost one-third of deaths in Brazil. Cardiovascular disease has become the leading cause of death in Brazil since 1960 due in part to poor eating habits, obesity, and insufficient physical activity. Consumption of high levels of sodium, added sugar, and saturated fat is a major driver of the development of cardiovascular disease. In this context, nutrition policies and interventions, such as the use of warning labels, are an important tool for reducing risk of diet-related diseases. The Brazilian Ministry of Health has recently announced efforts to combat the country's growing burden of diet-related noncommunicable diseases, and Brazil's National Health Surveillance Agency (ANVISA) has approved a more transparent and accessible system for communicating nutrition information for foods and beverages. The proposal will require labeling with a magnifying glass symbol on the front of products' packages to inform consumers about excess nutrients (i.e., sodium, sugar, saturated fat). Similar interventions have been implemented across Latin America, including Chile, Peru, and Mexico. A recent study in Chile demonstrated a reduction in purchases of food and drink items displaying warning labels.

This study seeks to test the effectiveness of different nutrient profiles to determine which products should carry the new labels in Brazil (i.e., the Pan-American Health Organization's profile or Brazil's National Health Surveillance Agency's proposed profile). Additionally, it seeks to assess whether the inclusion of information about products' ultra-processed nature further impacts consumers' product perceptions. The study will provide critical information for the Brazilian Ministry of Health on the effectiveness of the new label proposal and on strategies to inform Brazilians of product healthfulness.

Participants will be initially redirected from Cint (an online panel company). Following online consent and completion of a screening survey, participants will be redirected to an experimental online grocery store (Saruê), given a shopping list, and asked to shop for the items on the list as if in a real store. Upon redirection from Cint, participants will be randomly assigned into three arms: 1) control (no FOPLs); 2) FOPLs applied to products based on Brazil's National Health Surveillance Agency (ANVISA)'s nutrient profile model; or 3) front-of-package labels applied to products based on the Pan-American Health Organization (PAHO)'s nutrient profile model. After participants select products and check out, they will answer a survey about their perceptions about the labels and products carrying them. These questions will include self-reported responses to the content (e.g., elaboration, beliefs). After data collection, data on participants' selected products in the online grocery store will be analyzed to determine which nutrient profile was the most effective in decreasing participants' consumption of key nutrients.

Setting: The trial will take place in Saruê, an experimental online grocery store created for researchers to examine how front-of-package labels influence consumer purchases in a controlled but realistic environment. The online store reflects real-world prices and is modeled after Pão de Açúcar, a Brazilian online grocery store .

Recruitment: Participants will be recruited through Cint, a survey research firm. The eligibility criteria are residing in Brazil, being 18 years or older, and being responsible for at least half of the grocery shopping for one's household. Participants are ineligible if they were involved in any pre-testing related to the survey. Experiments conducted using online convenience samples, such as those recruited by Cint, largely replicate findings from studies conducted via probability-based samples. Cint will screen for eligibility and recruit participants from their pool of 8 million participants in Brazil. Approximately 3,000 participants will be recruited. As compensation, participants will receive incentives or points that can be redeemed for gift cards or goods per Cint's protocols.

Informed Consent: Participants will sign an informed consent form that follows a structure that is customary in Brazil.

Randomization: After the participant has signed the consent form, they will be randomly assigned to one of the three study arms. Randomization order will be determined a priori. Participants will have an equal chance of being randomized to each trial arm.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Resides in Brazil
* Does at least half of the grocery shopping for their household

Exclusion Criteria:

* Involved in any pre-testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3026 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Total sugar purchased | At completion of ~20 minute shopping task
  Total grams of sugar of products in a participant's shopping basket. This will be calculated by adding together the total sugar from each product in the participant's shopping basket. Sugar for each product will come from the product's nutrition facts panel. All products in the store are real life products that have designated nutrition facts panels.
Total saturated fat purchased | At completion of ~20 minute shopping task
  Total grams of saturated fat of products in a participant's shopping basket. This will be calculated by adding together the total saturated fat from each product in the participant's shopping basket. Saturated fat for each product will come from the product's nutrition facts panel. All products in the store are real life products that have designated nutrition facts panels.
Total sodium purchased | At completion of ~20 minute shopping task
  Total milligrams of sodium of products in a participant's shopping basket. This will be calculated by adding together the total sodium from each product in the participant's shopping basket. Sodium for each product will come from the product's nutrition facts panel. All products in the store are real life products that have designated nutrition facts panels.

SECONDARY OUTCOMES:
Percentage of ultra-processed products purchased | At completion of ~20 minute shopping task
  The percentage of products in a participant's shopping basket that are ultra-processed, as defined by the NOVA classification system.
Perceived healthfulness of unhealthy products | ~10 minute post-test computer survey following the ~20 minute shopping task
  Perceived healthfulness of sets of dairy products, bread, and chips with FOPLs according to study condition. Likert response options are on a 1 to 5 scale, with higher scores representing a higher perceived healthfulness of the products.
Perceived product appeal of unhealthy products | ~10 minute post-test computer survey following the ~20 minute shopping task
  Perceived product appeal of sets of dairy products, bread, and chips with FOPLs according to study condition. Likert response options are on a 1 to 5 scale, with higher scores representing a higher perceived product appeal of the products.
Health concerns of unhealthy products | ~10 minute post-test computer survey following the ~20 minute shopping task
  Perceived concern about health effects of sets of dairy products, bread, and chips with FOPLs according to study condition. Likert response options are on a 1 to 5 scale, with higher scores representing a higher health concern of the products.
Correct identification of high sugar/saturated fat/sodium content of unhealthy products | ~10 minute post-test computer survey following the ~20 minute shopping task
  Percentage of participants who correctly identified the sets of dairy products, bread, and chips as high in sugar, saturated fat, and/or sodium. Response options are yes, no, and I don't know.
Noticing of the label | ~10 minute post-test computer survey following the ~20 minute shopping task
  Percentage of participants who noticed the magnifying glass FOPLs in the experimental online grocery store. Response options are yes, no, and I don't know.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Clara Duran, PhD, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas, Campinas, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ribeiro AL, Duncan BB, Brant LC, Lotufo PA, Mill JG, Barreto SM. Cardiovascular Health in Brazil: Trends and Perspectives. Circulation. 2016 Jan 26;133(4):422-33. doi: 10.1161/CIRCULATIONAHA.114.008727. PMID 26811272
- [Background] World Health Organization. Noncommunicable Diseases (NCD) Country Profiles: Brazil. Published 2018. Accessed July 28, 2021. https://www.who.int/nmh/countries/bra_en.pdf.
- [Background] Wang YJ, Yeh TL, Shih MC, Tu YK, Chien KL. Dietary Sodium Intake and Risk of Cardiovascular Disease: A Systematic Review and Dose-Response Meta-Analysis. Nutrients. 2020 Sep 25;12(10):2934. doi: 10.3390/nu12102934. PMID 32992705
- [Background] Yang Q, Zhang Z, Gregg EW, Flanders WD, Merritt R, Hu FB. Added sugar intake and cardiovascular diseases mortality among US adults. JAMA Intern Med. 2014 Apr;174(4):516-24. doi: 10.1001/jamainternmed.2013.13563. PMID 24493081
- [Background] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300
- [Background] Agência Nacional de Vigilância Sanitária. Apresentação rotulagem nutricional_19a. Published 2020. Accessed July 28, 2021. https://www.gov.br/anvisa/pt-br/assuntos/noticias-anvisa/2020/aprovada-norma-sobre-rotulagem-nutricional/apresentacao-rotulagem-nutricional_19a.pdf/view
- [Background] Cancer Council Australia. Nutrient warning labels. Obesity Evidence Hub website. Published September 9, 2020. Accessed July 28, 2021. https://www.obesityevidencehub.org.au/collections/prevention/nutrient-warning-labels.
- [Background] Correa T, Fierro C, Reyes M, Dillman Carpentier FR, Taillie LS, Corvalan C. "Responses to the Chilean law of food labeling and advertising: exploring knowledge, perceptions and behaviors of mothers of young children". Int J Behav Nutr Phys Act. 2019 Feb 13;16(1):21. doi: 10.1186/s12966-019-0781-x. PMID 30760273

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT05789238/SAP_000.pdf